CLINICAL TRIAL: NCT04190576
Title: Subperiosteal Minimally Invasive Aesthetic Ridge Augmentation Technique With and Without Low Level Laser Therapy: A Comparative Clinical Trial
Brief Title: Minimally Invasive Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, PROFFESSOR, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_80831
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Alveolar Bone Loss; Bone Density Increased
MeSH Terms: conditions — Alveolar Bone Loss; Osteosclerosis | interventions — Low-Level Light Therapy; Bone Transplantation

STUDY DESIGN:
Intervention Model Description: Two groups were made one test and control. The control group were treated with MINIMALLY INVASIVE RIDGE AUGMENTATION technique alone and the test group were treated with adjunctive low-level laser therapy for bone regeneration.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minimally invasive ridge augmentation with LLLT (Experimental): Subperiosteal minimally invasive aesthetic ridge augmentation with G- Bone (Bone Graft) and low-level laser therapy
  Interventions: Device: Low Level Laser Therapy
- Minimally invasive ridge augmentation (Active Comparator): Subperiosteal minimally invasive aesthetic ridge augmentation with G- Bone (Bone Graft) alone
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Device: Low Level Laser Therapy — Hydroxyapatite bone graft with collagen
  Other Names: G- Bone (Bone Graft)

SUMMARY:
The present study is a human, prospective, randomised controlled clinical trial conducted to explore the outcome of a minimally invasive ridge augmentation technique with and without low level laser therapy. The trial is in accordance with the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010.

DETAILED DESCRIPTION:
Twenty healthy individuals satisfying the inclusion and exclusion criteria were recruited for the study. A detailed, thorough medical and dental history was obtained and each patient was subjected to comprehensive clinical and radiological examination. All patients were informed about the nature of the study, the surgical procedure involved, potential benefits and risks associated with the surgical procedure and written informed consent were obtained from all patients.

All the patients were treated with subperiosteal minimally invasive aesthetic ridge augmentation technique. the test group of ten were given low level laser therapy as an adjunct. The clinical and radiographic parameters were recorded at baseline and six months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple edentulous sites with Seibert's class 1 defects corresponding to colognes 1 and 2
* ASA 1 and 2
* Patients with an esthetic concern
* Good oral hygiene

Exclusion Criteria:

* Seibert's class 2 defects
* ASA 3 and 4
* Osteoporosis
* uncontrolled diabetes
* immunosuppression
* radiation therapy and bisphosphonate therapy
* Gingival thickness less than 2 mm

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Gain in Alveolar ridge width in millimeters | 6 months
  gain in alveolar ridge width at the agumented site in millimeters will be measured using Cone Beam Computed Tomography (CBCT) at baseline and six months

SECONDARY OUTCOMES:
Change in Bone density in Hounsefield's units | 6 months
  Change in Bone density in Hounsefield units will be measured using Cone Beam Computed Tomography (CBCT) at baseline and six months
Patient related outcomes of the surgical procedure in relation to 1) pain 2) discomfort and 3) swelling | one week
  Patient related outcomes during and after the procedure will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No